CLINICAL TRIAL: NCT05419843
Title: Up-front Matched Unrelated Donor Transplantation in Pediatric Patients With Idiopathic Aplastic Anemia: a Phase II Feasibility Study
Brief Title: Up-front Matched Unrelated Donor Transplantation in Pediatric Patients With Idiopathic Aplastic Anemia
Acronym: UPFRONT-MUD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP 200005
Record Dates: First submitted 2022-05-23; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Aplastic Anemia; Severe Aplastic Anemia; Moderate Aplastic Anemia Requiring Transfusions
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSCT arm group (Experimental): 1. Conditioning regimen
  2. Stem cell source Only Bone Marrow With a minimal target dose of 4x108 nucleated cells/kg recipient ideal body weight. If the graft is less rich than the minimum target dose, it can be administered at the discretion to the physician.
  3. GVHD Prophylaxis
  4. Prevention of EBV reactivation : Rituximab 150mg/m2 IV at Day+5 post HSCT.
  Interventions: Other: HSCT Arm group

INTERVENTIONS:
Other: HSCT Arm group — Conditioning regimen Stem cell source Only Bone Marrow With a minimal target dose of 4x108 nucleated cells/kg recipient ideal body weight. If the graft is less rich than the minimum target dose, it can be administered at the discretion to the physician.
  GVHD Prophylaxis Prevention of EBV reactivation : Rituximab 150mg/m2 IV at Day+5 post HSCT.

SUMMARY:
Pediatric patients with idiopathic aplastic anemia (AA) respond better than adults to immunosuppressive therapy (IST) but the long-term risks of relapse, ciclosporine dependence, and clonal evolution are high. UK investigators reported a 5-year estimated failure-free survival (FFS) after IST of 13.3%. In contrast, in 44 successive children who received a matched unrelated donor (MUD), hematopoietic stem cell transplantation (HSCT), there was an excellent estimated 5-year FFS of 95%. Forty of these children had previously failed IST. Because of those excellent results, up-front fully matched unrelated donor (MUD) hematopoietic stem cell transplantation (HSCT) became an attractive first-line option. In 2005 to 2014, a UK cohort of 29 children with idiopathic AA thus received MUD HSCTs as first-line therapy (they did not receive IST prior to HSCT). Results were excellent, with low Graft versus Host Disease rates and only 1 death (idiopathic pneumonia). This cohort was then compared with historical matched controls, transplanted or not. Outcomes for the up-front unrelated cohort HSCT were similar to Matched Related Donor HSCT and superior to IST and unrelated HSCT post-IST failure. Since then, many investigators are offering up-front MUD HSCT in pediatric patients worldwide. However, those results should be treated with extreme caution: 1) the design is retrospective; 2) the excellent up-front MUD HSCT may arise from the use of alemtuzumab in the conditioning regimen (alemtuzumab is not easily available worldwide) and 3) there was no formal quality-of-life assessment. Moreover, this strategy is highly dependent on donor identification (Caucasian patients have the highest likelihood of having a MUD) and donor not eventually receive HSCT because of the risk of infections/complications caused by unexpected donor delays or cancellation. Prospective trials are thus urgently needed to address the feasibility of such procedure, in term of timing (delay to offer MUD HSCT) and conditioning regimen (nothing is known of the use of other regimens, non alemtuzumab-based, in this setting).

The main objective of this Two-Stage Phase 2 multicenter study is to realize up-front HSCT within 2 months once a MUD has been identified.

ELIGIBILITY:
Inclusion Criteria:

* age<18years old
* Pediatric patients aged less than 18 years with idiopathic aplastic anemia and an indication for treatment (severe aplastic anemia or moderate aplastic anemia requiring transfusions)
* With a good probability to have a HLA-10/10 matched unrelated donor available (the patient needs to have at least 3 MUD identified within the book BMDW (Bone Marrow Donors Worldwide) or using the easy match software to be included)
* With usual criteria for allo-SCT:
* Lansky >70% for those below 16 years and Karnofsky > 70% for those above 16 years
* No severe and uncontrolled infection
* Adequate organ function: ASAT and ALAT ≤ 5N*, total bilirubin ≤ 2N, creatinine clearance > 70% of higher normal values for age.
* With health insurance coverage
* Contraception methods** for young girl and men of childbearing age must be prescribed during all the duration of the research.
* Parents having read and understand the information note and signed a written informed consent (the patient's agreement depending on his age will be sought)

  *because typical presentation of aplastic anemia post-hepatitis

  ** NB : The authorized contraceptive methods are:
* For women of childbearing age and in absence of permanent sterilization: oral, intravaginal or transdermal combined hormonal contraception, oral, injectable or transdermal progestogen-only hormonal contraception, intrauterine hormonal-releasing system (IUS).
* For man in absence of permanent sterilization: condoms

Exclusion Criteria:

Patients :

* With a matched related donor available
* With uncontrolled infection
* With seropositivity for HIV or HTLV-1 or active hepatitis B or C defined by a positive PCR HBV or HCV and associated hepatic cytolysis
* Renal failure with creatinine clearance below 70% of higher normal values for age
* Pregnant (βHCG positive) or breast-feeding
* With Heart failure according to NYHA (II or more)
* Preexisting acute hemorrhagic cystitis
* Urinary tract obstruction
* Yellow fever vaccine within 2 months before transplantation
* Who have any debilitating medical or psychiatric illness, which preclude understanding the inform consent as well as optimal treatment and follow-up (depending of his age and understanding).
* With Contraindication to treatments used during the research

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with upfront matched unrelated donor (MUD) hematopoietic stem cell transplantation (HSCT) effectively performed | within 2 months (60 days) after identification of a MUD
  Proportion of patients with upfront matched unrelated donor (MUD) hematopoietic stem cell transplantation (HSCT) effectively performed in the first two months after unrelated donor search.

SECONDARY OUTCOMES:
Graft failure incidence | up to 24 months
Neutrophils engraftment | at day 100
  Neutrophils engraftment will be defined as first day of 3 consecutive days with neutrophils >0.5 G/L
Platelets engraftment | at day 100
  Platelets engraftment will be defined as first day of 7 consecutive days with platelets >20 G/L
Absolute number of neutrophils | at 1 month
Absolute number of neutrophils | at 2 months
Absolute number of neutrophils | at 3 months
Absolute number of neutrophils | at 6 months
Absolute number of neutrophils | at 12 months
Absolute number of neutrophils | at day of last platelet and red blood cell transfusions (assessed up to 24 months)
Absolute numbers of platelets | at 1 month
Absolute numbers of platelets | at 2 months
Absolute numbers of platelets | at 3 months
Absolute numbers of platelets | at 6 months
Absolute numbers of platelets | at 12 months
Absolute numbers of platelets | up to 24 months
Acute GvHD incidence | at month 3
Chronic GvHD incidence | at 24 months
Relapse incidence | at 12 months
Relapse incidence | at 24 months
Progression free survival | at 12 months
Progression free survival | at 24 months
Incidence of CMV infection | at 12 months
Incidence of EBV infection | at 12 months
Incidence of severe infections | at 3 months
  Severe infections will be defined as CTACE grade 3-4
Incidence of severe infections | at 6 months
  Severe infections will be defined as CTACE grade 3-4
Incidence of severe infections | at 12 months
  Severe infections will be defined as CTACE grade 3-4
Incidence of severe infections | at 24 months
  Severe infections will be defined as CTACE grade 3-4
Non-relapse mortality | at 24 months
Overall survival | at 24 months
Quality of life questionnaires PedsQL | at inclusion
  Quality of life will be evaluated using PedsQL questionnaire. Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Quality of life questionnaires PedsQL | at 1 month
  Quality of life will be evaluated using PedQQL questionnaire.Higher scores associated with better health-related quality of life. Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Quality of life questionnaires PedsQL | at 3 months
  Quality of life will be evaluated using PedQQL questionnaire.Higher scores associated with better health-related quality of life. Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Quality of life questionnaires PedsQL | at 6 months
  Quality of life will be evaluated using PedsQL questionnaire. Higher scores associated with better health-related quality of life. Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Quality of life questionnaires PedsQL | at 12 months
  Quality of life will be evaluated using PedsQL questionnaire.Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Quality of life questionnaires PedsQL | at 24 months
  Quality of life will be evaluated using PedsQL questionnaire.Scores varies from 0 to100, with higher scores associated with better health-related quality of life.
Proportion of patients with a donor chimerism of 90% or more | at 1 month
Proportion of patients with a donor chimerism of 90% or more | at 3 months
Proportion of patients with a donor chimerism of 90% or more | at 6 months
Proportion of patients with a donor chimerism of 90% or more | at 12 months
Immune reconstitution | at 3 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL
Immune reconstitution | at 6 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL
Immune reconstitution | at 12 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Immune reconstitution | at 24 months
  Immune reconstitution will be done by analyzing T, B, NK, regulatory T cell levels in the peripheral blood. All have the same unit measure namely absolute numbers/microL.
Ferritin levels | at 3 months
Ferritin levels | at 6 months
Ferritin levels | at 12 months
Ferritin levels | at 24 months

IPD SHARING:
Plan to Share IPD: Undecided